CLINICAL TRIAL: NCT04326062
Title: Supporting Prescribing in Irish Primary Care: a Non-Randomised Pilot Study of a General Practice Pharmacist (GPP) Intervention to Optimise Prescribing in Primary Care
Brief Title: Supporting Prescribing in Irish Primary Care: General Practice Pharmacist Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Health Service Executive, Ireland (Other); University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Susan Smith, Prof Susan M Smith, Royal College of Surgeons, Ireland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GPP2071
Record Dates: First submitted 2018-04-26; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Polypharmacy; Multimorbidity
Keywords: Polypharmacy; Multimorbidity; General Practice; Pharmacist

STUDY DESIGN:
Intervention Model Description: Uncontrolled feasibility study based in general practices with a sub-set of patients completing a nested study collecting secondary patient reported outcome measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main Study (Experimental): A pharmacist will join the practice team for six months.
  Interventions: Other: Main Study
- PROM Study (Experimental): A nested Patient Reported Outcome Measure (PROM) study will be undertaken during month four and five of the six-month intervention period to explore the impact of the intervention in older adults (aged ≥65 years).
  Interventions: Other: PROM Study

INTERVENTIONS:
Other: Main Study — The pharmacist will participate in the management of repeat prescribing and undertake medication reviews (which will address high risk prescribing and potentially inappropriate prescribing, deprescribing and cost-effective and generic prescribing) with adult patients. Pharmacists will also provide prescribing advice regarding the use of preferred drugs, undertake clinical audits, join practice team meetings and facilitate practice-based education. Throughout the six-month intervention period, anonymised practice-level medication (e.g. medication changes) and cost data will be collected.
  Arms: Main Study
Other: PROM Study — For this, a sub-set of patients (n=200) aged ≥65 years on ≥10 repeat medicines will be recruited and invited to a medication review with the pharmacist. PROMs and healthcare utilisation data will be collected using patient questionnaires and a six-week follow-up review with these patients will also be conducted.
  Arms: PROM Study

SUMMARY:
The aim of this pilot study is to develop and test an intervention (defined as the General Practice Pharmacist [GPP] intervention) involving pharmacists working with General Practitioners (GPs) to optimise prescribing in Ireland. The study will determine the costs and potential effectiveness of the GPP intervention and, through engagement with key stakeholders, will explore the potential for an RCT of the GPP intervention in Irish general practice settings.

DETAILED DESCRIPTION:
Improving the quality and safety of prescribing for people with multiple chronic conditions and multiple medicines is a challenge for General Practitioners (GPs) and consequently, there has been an increased emphasis on ways to support GPs throughout this process. The integration of pharmacists into the general practice team is one approach being explored internationally and studies have shown that pharmacists, working as part of the general practice team, have influenced the safety and quality of prescribing. However, the evidence base is weak as there have been few high quality randomised controlled trials (RCTs) conducted and a range of modest effect sizes reported. Moreover, it is unclear whether such interventions can result in clinically significant improvements in patient outcomes. In Ireland, pharmacists are not integrated into general practice teams, therefore the feasibility of the integration of pharmacists into general practice warrants further exploration in the Irish primary care setting, prior to evaluation in a full scale RCT. The aim of this study is to develop and pilot test an intervention involving pharmacists, working within GP practices, to optimise prescribing in Ireland, which has a mixed public and private primary healthcare system.

ELIGIBILITY:
Inclusion Criteria for primary care practices:

* ≥1000 older patients (aged ≥65 years) on their patient panel.

Inclusion criteria for patients:

* Aged ≥65 years
* Taking ≥10 repeat medications
* Able to attend their primary care practice and participate in data collection.

Exclusion Criteria for patients:

* Psychiatric or psychological morbidity or cognitive impairment sufficient to impair the provision of informed consent
* Life-limiting illness likely to lead to death or major disability during the study follow-up period
* Patients who have already had a medication review/interacted with the pharmacist during the study period

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Changes in the number of medicines patients were prescribed. | Six months.
  We recorded the number of medicines that were stopped, started or changed as a result of the pharmacist doing a medication review.
Prevalence of potentially inappropriate prescribing. | Six months.
  We recorded the prevalence of potentially inappropriate prescribing identified by the pharmacist using validated indicators STOPP (Screening Tool of Older People' Prescriptions) and START (Screening Tool to Alert doctors to Right Treatment). STOPP and START are validated, explicit criteria used to identify potentially inappropriate prescribing in older people (those aged 65+ years).

SECONDARY OUTCOMES:
Patients' self-rated health-related quality of life. | Six months.
  We asked patients to rate their health-related quality of life using the European Quality of Life EQ5D-5L index score.
Self-rated attitudes of patients towards deprescribing of their medications. | Six months.
  We asked patients to rate their attitudes towards deprescribing of their medications using the revised Patients' attitudes towards deprescribing (rPATD) questionnaire.
Patients' self-rated treatment burden. | Six months.
  We asked patients to rate their experience of treatment burden using the Multimorbidity Treatment Burden Questionnaire (MTBQ).
Patients' self-rated beliefs about medicines | Six months.
  We asked patients to rate their beliefs about medicines using the Beliefs about Medicines Questionnaire.
Patients' self-rated health-related quality of life (VAS). | Six months.
  We asked patients to rate their health-related quality of life using the Visual Analogue Scale (range 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Smith, PhD, Principal Investigator — Royal College of Surgeons in Ireland
Locations (1):
- Royal College of Surgeons in Ireland, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Will be available from study PI on study completion
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication final papers
Access Criteria: Researchers requesting access to anonymised study data can contact the PI and access will be provided once all papers published from the study

REFERENCES:
- See also: Protocol for study — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-018-0311-7